CLINICAL TRIAL: NCT01113658
Title: Post-Market Clinical Evaluation of the Spiracur SNaP Wound Care System
Brief Title: Clinical Evaluation of the SNaP Wound Care System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated by Spiracur (original sponsor). Efforts were made to contact the PI/study team members, but were unsuccessful.
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNaP-113009
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Acute and Chronic Wounds; Pressure Ulcers; Trauma Wounds; Diabetic Foot Ulcers; Venous Stasis Ulcers
Keywords: negative pressure wound therapy; NPWT; Spiracur; SNaP Wound Care System
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNaP (Experimental): SNaP disposable, mechanically powered Negative Pressure Wound Therapy System
  Interventions: Device: SNaP Wound Care System

INTERVENTIONS:
Device: SNaP Wound Care System — The intervention is negative pressure wound therapy (NPWT) with the Spiracur SNaP Wound Care system for the treatment of a variety of acute and chronic wounds including pressure ulcers, trauma wounds, diabetic foot ulcers, venous stasis ulcers, and skin grafts.
  The Spiracur SNaP Wound Care system weighs less than 4 ounces, does not utilize an electric pump (device has no electrically powered parts), is fully disposable after use, and is designed for particularly small chronic wounds that require advanced wound care management. It delivers NPWT at a constant pressure level over several days without any required adjustments by the patient or clinician.
  Other Names: Spiracur SNaP Wound Care System; SNaP; The SNaP System

SUMMARY:
The purpose of this study is to assess the efficacy of design improvements of the Spiracur SNaP Wound Care System. This study prospectively evaluates the safety and efficacy of current and new design iterations of components of the FDA-cleared Spiracur SNaP Wound Care System in order to optimize safety, efficacy, and system performance.

ELIGIBILITY:
Inclusion Criteria:

* Wound < 10 cm in greatest diameter
* Patient >18 years of age
* Willing and able to sign informed consent

Exclusion Criteria:

* Patients with wound-related cellulitis
* Patients with thick eschar at wound base post debridement
* Patients with wounds located in an area not amenable to forming an air- tight seal
* Ulcers due to inflammatory conditions such as pyodermagangrenosum, rheumatoid arthritis, vasculitis, cryoglobulinemia, necrobiosislipoidicadiabeticorum, lupus or pancreatic panniculitis, cryofibrinogenemia, calcinosis cutis, scleroderma, Raynaud's syndrome
* Patient has untreated osteomyelitis
* Patient is allergic to wound care products
* Patient wounds with exposed blood vessels not suitable for negative pressure therapy
* Pregnant or pregnancy-suspected patients
* Subject actively participating in other clinical trials that conflict with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03 (Estimated); Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of complaints about device use and operation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristine K Nemes, DPM, Principal Investigator — Seton Hospital
Locations (2):
- United States (2):
  - San Francisco Center for Advanced Wound Care, Daly City, California
  - The SF Center For Advanced Wound Care At, Daly City, California